CLINICAL TRIAL: NCT02581774
Title: Management of Active Induction of Labor in Pregnancies Complicated With Oligohydramnios at Term; the Mode of Delivery and the Neonatal Outcomes
Brief Title: Active Induction of Labor in Pregnancies Complicated With Oligohydramnios at Term
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nazlı YENIGUL, MD, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 304
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2013-01

CONDITIONS: Oligohydramnios
Keywords: induction; cesarean delivery
MeSH Terms: conditions — Oligohydramnios

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- term isolated oligohydramnios: Labor Monitoring and normal delivery tracking
  Interventions: Other: normal delivery tracking
- prolonged pregnancies: Labor Monitoring and normal delivery tracking
  Interventions: Other: normal delivery tracking

INTERVENTIONS:
Other: normal delivery tracking — normal delivery tracking

SUMMARY:
The purpose of this study is to evaluate the risk of cesarean delivery in pregnancies complicated with isolated oligohydramnios managed by induction of labor. This prospective case-control study was conducted in Hamıdıye Sisli Etfal Teaching and Research Hospital between January 2013 and June 2014. 159 women with isolated oligohydramnios and 165 women with postdate pregnancies who met the inclusion criteria underwent induction of labor with dinoprostone or oxytocin. The rate and the indications of C/S deliveries were compared between two groups.

DETAILED DESCRIPTION:
The study was designed as a prospective study. The rates of cesarean section and maternal/fetal outcomes had been compared between pregnancies complicated with isolated oligohydramnios at term and postdate pregnancies. All patients with isolated oligohydramnios were term (37-40 weeks' gestation according to accurate last menstrual period and first trimester sonographic examination). Oligohydramnios was defined as an amniotic fluid index < 5 cm. The control group consisted of prolonged pregnancies in the absence of spontaneous labor and oligohydramnios. Prolonged pregnancy is diagnosed if 41 gestational weeks are completed according to accurate date of last menstrual period and first trimester ultrasound. All patients who accepted to join the study gave informed consent. All patients had a complete physical and obstetrical examination. Vital signs were recorded at regular intervals. The primary outcome measure was defined as cesarean section rates in pregnancies complicated with isolated oligohydramnios managed by induction of labor.

ELIGIBILITY:
Inclusion Criteria:

* term isolated oligohydramnios
* postdate pregnancies
* vertex presentation
* singleton pregnancies
* primigravid and multigravid women

Exclusion Criteria:

* women with presence of any chronic disease
* maternal condition complicating the pregnancy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients with isolated oligohydramnios were term (37-40 weeks' gestation according to accurate last menstrual period and first trimester sonographic examination). Oligohydramnios was defined as an amniotic fluid index < 5 cm. The control group consisted of prolonged pregnancies in the absence of spontaneous labor and oligohydramnios. Prolonged pregnancy is diagnosed if 41 gestational weeks are completed according to accurate date of last menstrual period and first trimester ultrasound.
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cesarean rates in pregnancies complicated with isolated oligohydramnios | up to 18 month

SECONDARY OUTCOMES:
Fetal distress rates | up to 18 month
Number of patients (fetus) with 5-min Apgar score < 7 | up to 18 month
Number of patients with meconium stained amniotic fluid | up to 18 month